CLINICAL TRIAL: NCT00856518
Title: Expiratory Muscle Training for Persons With Neurodegenerative Disease
Acronym: EMST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B6576-R
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Parkinson's Disease; Multiple Sclerosis
Keywords: Multiple Sclerosis; Parkinson's disease; Dysphagia
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: EMST (Active Comparator): The experimental group receives five weeks of expiratory muscle strength training (EMST) using a positive pressure threshold device
  Interventions: Device: EMST
- Arm 2: Sham group (Sham Comparator): The Sham group undergoes the same 5-week EMST exercise as the experimental group using the same device but without a spring for minimal pressure load
  Interventions: Device: Sham

INTERVENTIONS:
Device: EMST — Pressure threshold device (Expiratory Muscle Strength Trainer) targeted at increase muscle force generation of expiratory and submental muscles.
  Other Names: EMST 150
  Arms: Arm 1: EMST
Device: Sham — The same device just like the EMST but does not provide a load on the target muscle group
  Arms: Arm 2: Sham group

SUMMARY:
Respiratory difficulty is one of the primary factors leading to death in patients with Parkinson's Disease (PD) and Multiple Sclerosis. Both diseases are progressive degenerating diseases that cause difficulties in breathing, airway protection and swallowing. Patients with PD and MS typically become sedentary and lose endurance, maximal fitness levels and overall pulmonary function. Much of the research focus has been on the motor symptoms of PD and MS yet the pulmonary and swallowing complications are perhaps ultimately the most important disability as the diseases progress. The inability to generate adequate respiratory pressure is responsible for reduced cough magnitudes and cough response times. Cough is critical for the clearance of foreign materials in the airway helping to reduce infiltration of bacteria and subsequent respiratory infection. With reduced cough function an increased risk for pulmonary disease occurs due to a reduced ability to protect the airways. There are a number of promising outcomes from an expiratory strength-training program. By increasing expiratory muscle strength and expiratory pressure generation, effective breathing, clearance of the airway, and improved swallowing can occur. These explicit outcomes are predicted based on our experience with the use of an innovative device-driven, home-based expiratory strength training program focused on the expiratory muscles of respiration. This project focuses on following patients with PD and MS for an initial 5 weeks of strength training and them testing the outcome of a caregiver program for maintaining treatment effects.

DETAILED DESCRIPTION:
The proposed investigation will:

Determine if 5 weeks of Expiratory Muscle Strength Training (EMST) increases maximal expiratory driving pressure (MEP) and improves swallow, cough and breathing function in individuals with PD and MS. Following the post assessment of the 5 week EMST program we will then evaluate three different modules for monitoring the continuation of the treatment while assessing patient quality of life and caregiver burden/satisfaction. This will help us determine if one particular home training method results in different physiological and functional outcomes.

Aim 1. Determine the effects of an EMST program on swallow function, voluntary cough production and breathing function in individuals with PD and MS identified as below normal limits for their age and sex (via physiological measures).

Hypothesis 1: There will significant and positive treatment effects following 5 weeks of EMST on the measures of swallow, cough production and breathing function in those with PD and MS following 5 weeks of treatment.

Aim 2: Determine the outcome of three uniquely structured home treatment monitoring programs in maintaining the EMST post treatment effect for patients with MS and PD. These programs are referred to as: Education Module (A), Question Only (B), and Education Module plus Question (C). The monitoring system will be provided by VitelNet, a leading provider of home health monitoring, clinician-based telemedicine Hypothesis 2: Program C will provide greater maintenance of the EMST treatment effect for both patient groups compared to programs A and B.

Aim 3: Determine the effects of the home monitoring programs for improving patient quality of life and caregiver burden/satisfaction.

Hypothesis 3: Program C will provide greater improvements in patient quality of life and caregiver burden compared to programs A and B.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis Participants
* Diagnosis of primary, secondary, or relapsing-remitting MS by a neurologist
* Over 85% of the patient populations that come from the study sites demonstrate relapsing-remitting MS with an average relapse frequency of once every 3 years

Parkinson's Disease Participants

* Hoehn & Yahr, stage II and III as indicated by certified movement disorders neurologist

All Participants

* Between 35 and 80 years of age
* Non-smoking or no smoking within the previous five years
* No history of head and neck cancer, asthma or COPD, untreated hypertension
* Sufficient facial muscle strength so as to achieve and maintain adequate lip closure around a circular mouthpiece
* Cognition within normal limits as determined by the: Mini Mental Status Exam (MMSE; 1975No neurological (other than MS or PD) condition which adversely affects respiratory muscle or gas exchange system
* Reduced MEP's compared to published normative data for age and sex
* Reduced expiratory peak flow rates (6-8 L/s for young to middle age adults and 3.6 L/s for 65 and older) during voluntary cough production for age and sex (Bolser, personal communication; Smith-Hammond & Goldstein, 2006)
* Participant report of symptoms related to swallow impairment

Exclusion Criteria:

* DBS
* COPD
* Asthma
* Smoking or smoking within preceding 5 years

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis J. Daly, PhD MS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: EMST: Experimental Group
  Expiratory Muscle Strength Trainer: Pressure threshold device targeted at increase muscle force generation of expiratory and submental muscles.
- Arm 2: Sham Group: sham group
  sham device: Looks just like the EMST device but does not provide a load on the target muscle group
Period: Overall Study
Arm/Group | Arm 1: EMST | Arm 2: Sham Group
Started | 24 | 18
Completed | 20 | 16
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: EMST: Expiratory Muscle Strength Trainer: Pressure threshold device targeted at increase muscle force generation of expiratory and submental muscles.
- Arm 2: Sham Group: Sham Device: Looks just like the EMST device but does not provide a load on the target muscle group
- Total: Total of all reporting groups
Arm/Group | Arm 1: EMST | Arm 2: Sham Group | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9) | 58 (8) | 55 (9)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Expiratory Pressure (MEP)
Description: Expiratory pressure generating capacity assessed via handheld manometer.
Time Frame: at baseline and again after 5-week EMST exercise
Population: Out of the 42 recruited patients, 6 withdrew following the baseline MEP testing, citing travel or loss of interest as the reason. Therefore, 36 subjects were reported for the MEP test (n = 20 for EMST, n = 16 for sham).
Measure: Mean (Standard Deviation); unit: cm H2O
Groups:
- Arm 1: EMST: EMST Group
  Expiratory Muscle Strength Trainer: Pressure threshold device targeted at increase muscle force generation of expiratory and submental muscles.
- Arm 2: Sham: Sham group
  sham device: Looks just like the EMST device but does not provide a load on the target muscle group
Arm/Group | Arm 1: EMST | Arm 2: Sham
Number analyzed (Participants) | 20 | 16
cm H2O
  baseline | 78.6 (30.72) | 75.56 (27.68)
  post-training | 99.00 (32.97) | 99.38 (37.59)
Statistical Analysis 1: Comparison: Arm 1: EMST vs Arm 2: Sham; Test type: Superiority or Other; p = 0.899, Wilcoxon (Mann-Whitney) — EMST arm vs. Sham arm baseline MEP value comparison
Statistical Analysis 2: Comparison: Arm 1: EMST vs Arm 2: Sham; Test type: Superiority or Other; p = 0.946, Plum Ordinal Regression Test; EMST arm vs. Sham arm group comparison of treatment response
Statistical Analysis 3: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.00042, t-test, 2 sided; EMST arm post vs. pre-MEP comparison
Statistical Analysis 4: Comparison: Arm 2: Sham; Test type: Superiority or Other; p = 0.0019, t-test, 2 sided — Sham arm post vs. pre-MEP comparison

2. Primary Outcome: Penetration-Aspiration Scale Score
Description: The Penetration-Aspiration Scale (PAS) was used to measure swallow safety. PAS is an 8 point ordinal scale for quantification of penetration and aspiration. PAS measures the depth to which material enters the airway and if the material is expelled following penetration or aspiration. Categorical groupings of PAS scores include "normal to mild" (1-2), "moderate" (3-5) and "severe" (6-8, indicating that material has passed into the lower airway). These PAS scores may be useful in denoting clinically significant changes (e.g. moderate to mild) resulting from treatment or disease progression. The following table reports the percentage of participants (out of the respective total group participants in EMST and Sham) with changed PAS score of 1 point or more (improving or worsening) and without PAS score changes from pre- to post treatment. The data represent an exploratory quantification without statistical analysis.
Time Frame: at baseline and again after 5-week EMST exercise
Population: Out of the 42 recruited patients, 8 failed to complete the PAS test either at baseline or post training testing. Therefore, 34 subjects were reported for the PAS test (n = 20 for EMST, n = 14 for sham).
Measure: Number; unit: percentage of group participants
Arm/Group | Arm 1: EMST | Arm 2: Sham
Number analyzed (Participants) | 20 | 14
percentage of group participants
  with improved PAS after training | 40.0 | 14.3
  with unchanged PAS after training | 45.0 | 64.3
  with worsened PAS after training | 15.0 | 21.4

3. Primary Outcome: Swallow-related Quality of Life (SWAL-QOL)
Description: The SWAL-QOL is a validated and standardized tool that measures burden; symptom status including pharyngeal, oral, and saliva; fear; and mental health subdomains. Responses are determined according to an ordinal scale where 1 equals a severe problem and 5 equals no problem. The SWAL-QOL provides an overall score as well as subscale scores. Subjects rate quality of life as follows (expressed as percentage of the possible perfect score): little to no impact (81% - 100%), mild impact (61% - 80%), moderate impact (41% - 60%), severe impact (21% - 40%), and profound impact (0% - 20%).
Time Frame: at baseline and after 5-week of EMST exercise
Population: Out of the total 42 recruited study participants, ten either did not show up for the SWAL-QOL test or only partially answered the questionnaire. Thus, 32 remaining participants (n = 19 for EMST, and n = 13 for Sham) were reported.
Measure: Mean (Standard Deviation); unit: percentage of possible perfect score
Arm/Group | Arm 1: EMST | Arm 2: Sham Group
Number analyzed (Participants) | 19 | 13
percentage of possible perfect score
  pre-training total SWAL-QOL | 83.3 (11.5) | 81.4 (10.9)
  post-traing total SWAL-QOL | 88.1 (10.8) | 84.4 (8.5)
  pre-training Burden | 90.0 (20.0) | 80.8 (25.0)
  post-training Burden | 97.4 (7.3) | 86.2 (18.9)
  pre-training Pharyngeal | 73.5 (16.9) | 75.4 (13.0)
  post-training Pharyngeal | 82.4 (16.6) | 77.6 (11.6)
  pre-training Saliva | 84.2 (16.2) | 83.1 (13.5)
  post-training Saliva | 92.3 (9.5) | 83.6 (15.8)
  pre-training Oral | 95.3 (7.0) | 91.2 (13.1)
  post-training Oral | 96.9 (4.5) | 91.2 (9.8)
  pre-training Fear | 80.5 (22.2) | 79.2 (14.8)
  post-training Fear | 89.2 (20.4) | 84.6 (11.3)
  pre-training Mental Health | 87.2 (21.5) | 83.4 (16.5)
  post-training Mental Health | 94.1 (18.2) | 90.2 (13.0)
Statistical Analysis 1: Comparison: Arm 1: EMST vs Arm 2: Sham Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — EMST arm vs. Sham arm baseline total score and subscale score comparison
Statistical Analysis 2: Comparison: Arm 1: EMST vs Arm 2: Sham Group; Test type: Superiority or Other; p > 0.05, Plum Ordinal Regression Test; EMST arm vs. Sham arm group comparison of treatment response for total score and all subscale scores except for Burden and Pharyngeal domains
Statistical Analysis 3: Comparison: Arm 1: EMST vs Arm 2: Sham Group; Test type: Superiority or Other; p = 0.014, Plum Ordinal Regression Test; EMST arm vs. Sham arm group comparison of treatment response in Burden domain
Statistical Analysis 4: Comparison: Arm 1: EMST vs Arm 2: Sham Group; Test type: Superiority or Other; p = 0.022, Plum Ordinal Regression test; EMST arm vs. Sham arm group comparison of treatment response in Pharyngeal domain
Statistical Analysis 5: Comparison: Arm 2: Sham Group; Test type: Superiority or Other; p > 0.05, Wilcoxon Signed Ranks Test — Sham arm post vs. pre-treatment comparison for the total SWAL-QOL score and subscale scores except for the Burden and Mental Health domains
Statistical Analysis 6: Comparison: Arm 2: Sham Group; Test type: Superiority or Other; p = 0.038, Wilcoxon Signed Ranks Test; Sham arm post vs. pre-treatment comparison in Burden domain
Statistical Analysis 7: Comparison: Arm 2: Sham Group; Test type: Superiority or Other; p = 0.031, Wilcoxon Signed Ranks Test; Sham arm post vs. pre-treatment comparison in Mental Health domain
Statistical Analysis 8: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.027, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Burden domain
Statistical Analysis 9: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.016, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Mental Health domain
Statistical Analysis 10: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.007, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Pharyngeal domain
Statistical Analysis 11: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.036, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Saliva domain
Statistical Analysis 12: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.004, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Fear domain
Statistical Analysis 13: Comparison: Arm 1: EMST; Test type: Superiority or Other; p = 0.016, Wilcoxon Signed Ranks Test; EMST arm post vs. pre-treatment comparison in Total SWAL-QOL score

ADVERSE EVENTS:
Time Frame: Seven-week period (baseline testing at week 1, then 5 weeks of the experimental training, and post-training testing at week 7)
Arm/Group | Arm 1: EMST | Arm 2: Sham Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 0/24 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes